CLINICAL TRIAL: NCT06465238
Title: A Phase II Study of the Efficacy and Safety of SHR-A1921 or SHR-A2009 in Patients With Previously Treated Advanced NSCLC
Brief Title: Clinical Study of SHR-A1921 or SHR-A2009 in Previously Treated Advanced NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, Professor, Henan Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-IIT-SHRA2009-SHRA1921
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group 1 (Experimental): SHR-A2009
  Interventions: Drug: SHR-A2009
- Treatment group 2 (Experimental): SHR-A1921
  Interventions: Drug: SHR-A1921

INTERVENTIONS:
Drug: SHR-A2009 — Treatment group: Subjects will receive an intravenous infusion of SHR-A2009 until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the study.
  Arms: Treatment group 1
Drug: SHR-A1921 — Treatment group: Subjects will receive an intravenous infusion of SHR-A1921 until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the study.
  Arms: Treatment group 2

SUMMARY:
This study is an open-label Phase II clinical trial to evaluate the safety and efficacy of SHR-A1921 or SHR-A2009 in patients with advanced NSCLC who progressed after standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent;
2. Aged 18-75 years (inclusive), males and females;
3. Has a histologically or cytologically confirmed diagnosis of metastatic NSCLC (according to 8th AJCC/UICC Classification);
4. Has failed to standard therapy and disease progressed after antibody-conjugated drugs therapy;
5. Has at least 1 measurable lesion per RECIST 1.1;
6. Patients with ECOG score of 0-1;
7. Life expectancy ≥12 weeks;
8. Have adequate organ function;
9. Participants agrees to use contraception, and be abstinent from heterosexual intercourse during the treatment period and for ≥180 days after the last dose of study treatment.

Exclusion Criteria:

1. Histologically or cytologically confirmed presence of small-cell lung cancer or other benefit-limiting tumor components;
2. Untreated brain metastasis or accompanied by meningeal metastases, spinal cord compression;
3. Cancerous ascites, pleural effusion or pericardial effusion with clinical symptoms;
4. Subjects who have received systemic anti-tumor treatments prior to the initiation of the study treatment;
5. Has received major organ surgery or high-intensity thoracic radiotherapy within before first dose of study therapy；
6. Has a history of a second malignancy;
7. Has a history of non-infectious ILD/pneumonitis that required steroids, or has current ILD/pneumonitis;
8. Subjects with active pulmonary tuberculosis infection；
9. Serious infection before the first dose；
10. Uncontrolled cardiac diseases or symptoms;
11. Arterial/venous thrombosis events occurred before the first dose；
12. Hypertension that can not be well controlled through antihypertensive drugs，previous hypertensive crisis or hypertensive encephalopathy；
13. Has a history of active chronic enteritis;
14. Has a history of bleeding prior to the initiation of the study treatment;
15. History of immunodeficiency disease or organ transplant;
16. Subjects with active hepatitis B or active hepatitis C;
17. Has unresolved toxicities from previous anticancer therapy;
18. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients of SHR-A1921or SHR-A2009;
19. Subjects with other potential factors that may affect the study results or result in the premature discontinuation as determined by the investigator, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, or family or social factors that could affect the safety of the patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 12 months
  Assessed by Investigator According to RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
  Assessed by Investigator According to RECIST v1.1
overall survival (OS) | up to 24 months
  OS is the time from the date of first dose until the date of death by any cause.
Duration of response(DoR ) | up to 12 months
  Assessed by Investigator According to RECIST v1.1
Disease control rate (DCR) | up to 12 months
  Assessed by Investigator According to RECIST v1.1
Time to Response (TTR) | up to 12 months
  Assessed by Investigator According to RECIST v1.1
The incidence and severity of adverse events (AEs) | from Day1 to 90 days after last dose
  Rated based on CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No